CLINICAL TRIAL: NCT03282032
Title: Preconditioning of One-lung Ventilation for Lung Protection
Brief Title: Preconditioning of One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JHSeo_preconditioning
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-08

CONDITIONS: One Lung Ventilation
MeSH Terms: interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-lung ventilation (Experimental): Before surgical incision, 2-min of OLV followed by 2-min of TLV (1 cycle) is performed for 5 cycles.
  Interventions: Other: One-lung ventilation
- Two-lung ventilation (No Intervention): Maintain two-lung ventilation until surgical incision

INTERVENTIONS:
Other: One-lung ventilation — The patient undergoing thoracic surgery is intubated with double lumen tube after induction of general anesthesia with propofol and remifentanil.
  In the intervention group, 5 cycles of one-lung ventilation preconditioning (2-min of one-lung ventilation and 2-min of two-lung ventilation for 1 cycle) is performed before surgical incision. One-lung ventilation is done at dependent lung with FiO2 100% and tidal volume 6 ml kg-1. Two-lung ventilation is done with FiO2 50%, tidal volume 8 ml kg-1.
  Other Names: Preconditioning
  Arms: One-lung ventilation

SUMMARY:
To observe the effect of one-lung ventilation (OLV) preconditioning on perioperative oxygenation during thoracic surgery.

DETAILED DESCRIPTION:
For lung isolation and better surgical view, one-lung ventilation(OLV) is essential for thoracic surgery. However, OLV may cause serious pulmonary complications due to intraoperative hypoxia.

Animal studies showed a positive effect of OLV preconditioning (Intermittent OLV before surgical intervention) on perioperative pulmonary oxygenation.

Thus, we designed a study to observe the effect of OLV preconditioning on perioperative oxygenation during thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracic surgery which requires one-lung ventilation with lateral decubitus position

Exclusion Criteria:

* Patients with severe cardiopulmonary disease, COPD, previous surgical history of pulmonary disease
* Thoracic surgery for pneumonectomy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxemia | during one-lung ventilation, up to 5 hours
  SpO2 < 95%
P/F ratio | 30min after surgical incision
  PaO2/FIO2 ratio

SECONDARY OUTCOMES:
Pulmonary complications | 6, 24, 48 hours after surgery, during hospital stay.
  Acute lung injury, acute respiratory distress syndrome, atelectasis, pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Benumof JL. Intermittent hypoxia increases lobar hypoxic pulmonary vasoconstriction. Anesthesiology. 1983 May;58(5):399-404. doi: 10.1097/00000542-198305000-00001. PMID 6837992